CLINICAL TRIAL: NCT00003231
Title: Preoperative Chemotherapy in Non-Small Cell Lung Cancer (NSCLC) Patients With Mediastinal Lymph Node Metastases (Stage IIIA, N2)
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SAKK 16/96; SWS-SAKK-16/96; EU-97034
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Docetaxel; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with docetaxel and cisplatin followed by surgery in treating patients with stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and toxic effects of docetaxel plus cisplatin in patients with stage IIIA non-small cell lung cancer. II. Assess the clinical and pathological response rate to this therapy in this patient population. III. Compare the benefit of surgery in terms of overall survival of responding and nonresponding patients.

OUTLINE: Patients receive infusions of docetaxel over 1 hour on day 1, followed by infusions of cisplatin over 1 hour on days 1-2. Treatment is repeated for three 21 day courses. Patients undergo tumor resection and mediastinal lymph node dissection. Patients are to receive postoperative radiotherapy within 4 weeks of resection if the tumor reaches the resection margins and/or the first mediastinal lymph node levels are involved. Patients will be followed until death.

PROJECTED ACCRUAL: Approximately 5-40 patients will be accrued within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IIIA non-small cell lung cancer (NSCLC)(including squamous, adenocarcinoma, large cell, and poorly differentiated NSCLC) Nodal metastases of T1-3 N2 M0 No distant metastases

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance Status: WHO 0-2 Life Expectancy: Not specified Hematopoietic: Leucocytes greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin within normal limits AST or ALT no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine clearance greater than 60 mL/min No hypercalcemia Cardiovascular: No unstable cardiac disease No congestive heart failure No angina pectoris No significant arrhythmias No prior history of myocardial infarction within 3 months Pulmonary: Lung function test with a forced expiratory volume greater than 1.2 L/sec Neurologic: No dementia No peripheral neuropathy greater than grade 1 No psychosis No seizure disorders Other: No prior or concurrent malignancies, except: Nonmelanoma skin cancer Carcinoma in situ of the cervix No active uncontrolled infection or other serious medical conditions No diabetes mellitus treated with insulin No gastric ulcers

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: No prior corticosteroids or other endocrine therapy No concurrent treatment with prednisone (except for prophylaxis, treatment of acute hypersensitivity, or chronic treatment initiated greater than 6 months prior to study entry) Radiotherapy: No prior radiotherapy Surgery: No prior surgery for malignancy Other: No concurrent treatment with other experimental drugs No involvement in clinical trials within 30 days of study No prior treatment with other cytostatic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1997-04; Primary Completion 2000-09 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Betticher, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (9):
- Switzerland (9):
  - Kantonspital Aarau, Aarau
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Betticher DC, Hsu Schmitz SF, Totsch M, Hansen E, Joss C, von Briel C, Schmid RA, Pless M, Habicht J, Roth AD, Spiliopoulos A, Stahel R, Weder W, Stupp R, Egli F, Furrer M, Honegger H, Wernli M, Cerny T, Ris HB; Swiss Group for Clinical Cancer Research (SAKK). Prognostic factors affecting long-term outcomes in patients with resected stage IIIA pN2 non-small-cell lung cancer: 5-year follow-up of a phase II study. Br J Cancer. 2006 Apr 24;94(8):1099-106. doi: 10.1038/sj.bjc.6603075. PMID 16622435
- [Result] Betticher D, Hsu Schmitz S, Roth A, et al.: Neoadjuvant therapy with docetaxel and cisplatin in patients with non-small cell lung cancer (NSCLC), stage IIIA, pN2: a large phase II study with 59 months of follow-up. [Abstract] Lung Cancer 50 (Suppl 2): A-O-032, S14, 2005.
- [Result] Betticher DC, Hsu Schmitz SF, Totsch M, Hansen E, Joss C, von Briel C, Schmid RA, Pless M, Habicht J, Roth AD, Spiliopoulos A, Stahel R, Weder W, Stupp R, Egli F, Furrer M, Honegger H, Wernli M, Cerny T, Ris HB. Mediastinal lymph node clearance after docetaxel-cisplatin neoadjuvant chemotherapy is prognostic of survival in patients with stage IIIA pN2 non-small-cell lung cancer: a multicenter phase II trial. J Clin Oncol. 2003 May 1;21(9):1752-9. doi: 10.1200/JCO.2003.11.040. PMID 12721251
- [Result] Fruh M, Betticher DC, Stupp R, Xyrafas A, Peters S, Ris HB, Mirimanoff RO, Ochsenbein AF, Schmid R, Matzinger O, Stahel RA, Weder W, Guckenberger M, Rothschild SI, Lardinois D, Mach N, Mark M, Gautschi O, Thierstein S, Biaggi Rudolf C, Pless M; Swiss Group for Clinical Cancer Research (SAKK). Multimodal Treatment in Operable Stage III NSCLC: A Pooled Analysis on Long-Term Results of Three SAKK trials (SAKK 16/96, 16/00, and 16/01). J Thorac Oncol. 2019 Jan;14(1):115-123. doi: 10.1016/j.jtho.2018.09.011. Epub 2018 Sep 26. PMID 30267838